CLINICAL TRIAL: NCT04406363
Title: Confinement Effect on Low Back Pain Intensity in Chronic Low Back Pain Patients
Acronym: CONFI-LOMB
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: CONFI-LOMB
Record Dates: First submitted 2020-05-06; First posted 2020-05-28 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Chronic Low-back Pain
Keywords: confinement; chronic low back pain; changes in pain intensity; bio-psycho-social and occupational factors; physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: non interventional — non interventional

SUMMARY:
The current situation, linked to the pandemic of the new coronavirus SARS-CoV-2 generates health concerns, but is also accompanied by many other psychological, social, economic, professional, etc. consequences as well as numerous changes in behavior and lifestyles, notably due to confinement.

While the prevention of chronic low back pain and its management are primarily based on the practice of regular physical and sports activity, other psychological factors (stress, anxiety, depression), socioeconomic (low level of education, resources), professionals (physical workload, job dissatisfaction), etc. also have a major role in the onset and the persitence of low back pain.

Thus, it is to be supposed that the current context, and more particularly the confinement to which the population has been constrained for almost 2 months, have and will have notable consequences on the evolution of lumbar symptoms in chronic low back pain patients. However, the entanglement of different factors related to containment will potentially have different consequences depending on the individual. It therefore seems difficult to predict how the lumbar symptoms will develop in this population. Indeed, if it can imagined that the decrease in regular physical activity and the increase in anxiety in this context of insecurity could lead to an increase in pain, it could just as well consider that the decrease in stress work, strenuous physical work or travel time from work to home can, on the contrary, have a favorable effect.

The objective of this study is to assess the confinement effect on low back pain intensity in chronic low back pain patients.

This is an observational, descriptive, transversal and pluricentric study conducted by a single questionnaire.

DETAILED DESCRIPTION:
Patients who consulted one of the study investigators (rheumatologist and algologist) for the management of a common chronic low back pain between January 1, 2020 and March 17, 2020 (begining of the French confinement) and who meet inclusion criteria will be offered to participate to the study.

Eligible subjets will be preselected by the study investigators (from the medical file). The initial solicitation of a potential subject will be made by a phone contact by the investigator who treat him/her for his chronic low back pain. Subjects who agree to participate in the study will be offered to respond to a questionnaire by phone.

The questionnaire (no more than 10 minutes) will assess the sociodemographic status, the confinement conditions, the new coranavirus infection status, changes in low back pain intensity during the confinement, incapacity related to low back pain, physical activities practice before and during the confinement, anxiety and depression, continuation of occupational activity and teleworking practice during the confienment .

The main objective of this study is to assess the impact of confinement on change in low back pain intensity. The main endpoint is the proportion of subjects with a significant change in their low back pain during confinement, defined by the items "much worse" and "moderately worse", or "much improved" and "moderately improved" respectively.

The secondary objectives are to assess:

1. the association between the conditions of confinement and low back pain intensity;
2. the association between the confinement conditions and disability related to low back pain;
3. the association between infection with the new SARS-CoV-2 coronavirus and change in low back pain intensity;
4. the association between the confinement conditions and the quality of life as well as the state of psychological health;
5. the impact of confinement on the use of care and the consumption of medication and psychoactive substances for low back pain;
6. the association between working conditions and / or teleworking and the low back pain intensity;
7. the association between socio-economic factors and modalities as well as the experience of confinement.

Given the exploratory nature of this study, the required number of subjects is empirically estimated at 350 subjects in total.

Qualitative and quantitative data will be described (averages or percentages). A chi² test will be performed to compare the percentages between the different subgroups studied. A Student test will be carried out to compare the means between the different subgroups studied. An alpha risk of less than 5% will be considered significant.

For each of the parameters of interest studied, the bivariate analysis may be supplemented by a multivariate analysis adapted to the criterion to be explained if the conditions of validity of this multivariate analysis are met.

ELIGIBILITY:
Inclusion Criteria:

* Major patients (men and women) with common chronic low back pain (i.e. without identified underlying cause)
* Patients who benefited from a consultation with a specialist doctor (rheumatologist or algologist) from the recruitment centers for common chronic low back pain between January 1, 2020 and March 17, 2020 (begining of the French confinement) included
* Patients who received information with non-opposition

Exclusion Criteria:

* Pain other than spinal pain not allowing to discriminate low back pain (fibromyalgia, chronic pain syndrome, etc.)
* Low back pain of secondary origin (infectious, tumor, fracture, inflammatory, etc.)
* Comorbidities limiting the practice of physical and sporting activities (severe heart or respiratory failure, arteriopathy of the lower limbs with lameness, etc.)
* Poor understanding of the French language
* Pregnant, lactating or parturient women
* Vulnerable adults within the meaning of the law
* Person deprived of their liberty by judicial or administrative decision
* Person under psychiatric care under duress
* Person admitted to a health or social establishment for purposes other than that of research
* Person subject to a legal protection measure
* Person out of state to express consent
* Person opposed to participating in the research

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who consulted one of the study inestigators (rheumatologist or algologist) for the management of common chronic low back pain between January 1, 2020 and March 17, 2020 inclusive and who meet the inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-06-02 (Estimated); Primary Completion 2020-06-02 (Estimated); Study Completion 2020-06-21 (Estimated)

PRIMARY OUTCOMES:
Impact of confinement on the low back pain intensity | at inclusion
  Proportion of subjects having a significant change in their low back pain intensity during confinement, defined by the items "much worse" and "moderately worse", or "much improved" and "moderately improved" respectively.The meaning of this significant change (worsening or improvement) will also be described.

SECONDARY OUTCOMES:
Correlation between confinement conditions and low back pain intensity | at inclusion
  Change in low back pain intensity between before and during confinement evaluated by a numerical pain scale rated from 0 to 10 (0 = no pain ; 10 = worst imaginable pain). Confinement conditions (alone or in a group, space, etc.) and the practice of physical and sporting activities during confinement (weekly duration, etc.)
Correlation between confinement conditions and disability related to low back pain | at inclusion
  Disability measured by the "incapacity" sub-score of the "Core Outcome Measures Index" (COMI) questionnaire
Correlation between infection with the new SARS-CoV-2 coronavirus and change in low back pain intensity | at inclusion
  Occurrence of a SARS-CoV-2 infection and its level of severity (confirmed diagnosis, few or no symptoms, symptoms severely limiting daily activities, hospitalization in a conventional service or in intensive care)
Correlation between confinement conditions and quality of life as well as psychological health | at inclusion
  Quality of life and levels of anxiety and depression evaluated with the COMI-AD sub-score (modified version of the COMI integrating the state of psychological health);
Impact of confinement on the use of care and the consumption of medication and psychoactive substances for low back pain | at inclusion
  Use of care, drug consumption and psychoactive substances (tobacco, cannabis, alcohol, anxiolytics) for low back pain
Correlation between working conditions and / or teleworking and low back pain intensity | at inclusion
  Modalities of the the ocupational activity continuation (continuation of the activity, evolution of the working time, telework and modalities of establishment)
Correlation between socio-economic factors and modalities as well as the experience of confinement | at inclusion
  Experience of confinement. Socio-economic characteristics of the participants (age, sex, department, job and socio-professional category).

CONTACTS AND LOCATIONS:
Locations (1):
- Petit, Angers, France

IPD SHARING:
Plan to Share IPD: No